CLINICAL TRIAL: NCT04176055
Title: Prospective Evaluation of Symptoms and Open Label Haloperidol in Cannabinoid Hyperemesis Syndrome (HALO)
Brief Title: Treatment Strategies in CHS
Acronym: HALO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Christopher Andrews, Principal Investigator, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB19-1197
Record Dates: First submitted 2019-11-20; First posted 2019-11-25 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Cannabis Hyperemesis Syndrome
MeSH Terms: conditions — Cannabinoid Hyperemesis Syndrome | interventions — Haloperidol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HALO (Experimental)
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Haloperidol — haloperidol intervention

SUMMARY:
Background:

In the gastrointestinal (GI) system, the most well-described manifestation of prolonged cannabis use is cannabinoid hyperemesis syndrome (CHS). CHS is characterized by severe cyclic nausea and vomiting and associated with abdominal pain.Currently, the generally accepted management for CHS is complete cannabis abstinence as traditional anti-emetics appear to be minimally effective. Preliminary reports from emergency departments suggest that intravenous haloperidol, a typical anti- psychotic, provides effective symptomatic relief in CHS.

Objective:

1. To learn more about how cannabis use relates to the management of CHS.
2. To learn if haloperidol is effective in treating the symptoms of CHS.

Eligibility:

Alberta residents with ongoing cannabis use, who have completed the baseline study, are ≥ 18 years and ≤ 65 years, and have gastrointestinal symptomology as measured by GCSI > 2 or PAGI-SYM > 2 (upper or lower abdominal pain subscale).

Design:

Participants will answer a series of questionnaires online. Study specific questions relating to symptoms, cannabis use, and anxiety and depression will be administered. Confirmation of cannabis cessation will be assessed with urine creatinine and cannabis metabolite measures. Salivary cortisol will be used to asses the stress response.

DETAILED DESCRIPTION:
In the gastrointestinal (GI) system, the most well-described manifestation of prolonged cannabis use is cannabinoid hyperemesis syndrome (CHS). CHS is characterized by severe cyclic nausea and vomiting and associated with abdominal pain.The pathophysiology of CHS is poorly understood but may involve alterations gut motility and/or activation of the hypothalamic-pituitary-adrenal (HPA) axis.

Our endogenous endocannabinoid system contains the cannabinoid receptor type I (CB1) and type II (CB2), and their ligands, anandamide (AEA) and 2-arachidonylglycerol (2-AG). CB1 receptors are widely distributed throughout the central and peripheral nervous system, including the myenteric plexus of the GI tract. In humans, oral Δ9-THC (an active cannabis compound) reduces gastric emptying and patients with slow transit constipation have increased expression of endogenous endocannabinoids and higher CB1 receptor expression. In CHS, chronic cannabis use may cause significant activation of peripheral, gut-located CB1.

The hypothalamic-pituitary- adrenal (HPA) axis, the main neuroendocrine system activated in response to stressful stimuli may also be involved in CHS. Activation of centrally located CB1 receptors by 2-AG plays a crucial role in down-regulating the HPA axis in recovery from stress. Reduction in 2-AG activity within the hypothalamus by stress, leads to reduced hypothalamic CB1 receptor activation; this reduced CB1 activation is also observed in prolonged cannabis use.

Currently, the generally accepted management for CHS is complete cannabis abstinence as traditional anti-emetics appear to be minimally effective.Preliminary reports from emergency departments suggest that intravenous haloperidol, a typical anti- psychotic, provides effective symptomatic relief and has become a first-line agent for acute CHS.

Outcome measures:

The primary endpoints will look at the correlation between quantitative weekly cannabis use and gastrointestinal symptoms at week 8 and the mean change of the GI symptoms from week 8 to week 12 during.

ELIGIBILITY:
Inclusion Criteria:

1. Completed Baseline study prior to enrollment
2. Age ≥ 18 years and ≤ 65 years
3. Gastrointestinal symptomology as measured by GCSI > 2 or PAGI-SYM > 2 (upper or lower abdominal pain subscale)
4. Ongoing cannabis use (> 1g/wk)
5. Resident of Alberta with valid Alberta Health Care number

Exclusion Criteria:

1. Pregnancy and/or breastfeeding
2. Corrected QT interval measured on ECG > 450 ms for males or >470 ms for females
3. History of seizure, venous thromboembolism (VTE), psychosis, Parkinson's disease or spastic disorder
4. Concurrent diagnosis of or suspected gastroparesis or functional dyspepsia
5. Diabetes with neuropathy.
6. Any gastrointestinal, neurological, or other illness felt by the investigators to be potentially involved in symptom generation or pose a safety risk to inclusion in this study.
7. Previous gastric or intestinal surgery which may lead to symptoms
8. Use of concomitant medications which cannot be stopped for the 4-week haloperidol phase of the study: including narcotics, antihistamines such as diphenhydramine (Benadryl) or dimenhydrinate (Gravol), dopamine antagonists (domperidone, metoclopramide, risperidone, clozapine, quetiapine), macrolide antibiotics, prokinetics (prucalopride), tricyclic antidepressants (TCA) at doses >50 mg, barbiturates, 5HT3 antagonists (ondansetron).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Correlation between quantitative weekly cannabis use and GI symptoms at week 8 | 1st 8 weeks of the 12 week study for outcome 1
  GI symptoms will be measured PAGI-SYM, a 20-item Likert-type measure with six sub classes. Cannabis use will be measured by the cannabis consumption inventory (DFAQ-CU).The participants will fill out the questionnaires every 2 weeks.
Mean change in GI symptoms from week 8 to week 12 | final 4 weeks of the 12 week study for outcome 2
  GI symptoms will be measured PAGI-SYM, a 20-item Likert-type measure with six sub classes. The participants will fill out the questionnaire every 2 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada